CLINICAL TRIAL: NCT05250882
Title: Enhanced Perioperative Care for Improving Outcomes After Colorectal Resection by Implementation of Best Practice for the Prevention of Anastomotic Leakage - Double Check Study: Protocol for a Multicenter Open-label Trial
Brief Title: Enhanced Perioperative Care for the Prevention of Colorectal Anastomotic Leakage
Acronym: DOUBLE CHECK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Freek Daams, Principal Investigator, Gastrointestinal Surgeon, Amsterdam UMC, location VUmc
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020.0634
Record Dates: First submitted 2022-01-20; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Anastomotic Leak Small Intestine; Anastomotic Leak Large Intestine; Anastomotic Leak Rectum; Intraoperative Awareness
Keywords: Riskfactor; Colorectal resection; Intraoperative condition; Perioperative care
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Intervention Model Description: Open label multicenter trial with historic controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double Check enhanced perioperative care protocol (Experimental): Perioperative care according to a best practice protocol focussing on optimizing the intraoperative condition of the patient and thereby minimalize exposure to 6 known modifiable independent intraoperative risk factors: anemia, hypothermia, epidural anesthesia, vasopressor drug administration, incorrect antibiotic prophylaxis and hyperglycemia.
  Interventions: Other: Enhanced perioperative care protocol
- Current practice (No Intervention): Perioperative care according to usual practice. Historical controls from the previously conducted LekCheck study will be used as replacement of a control arm.

INTERVENTIONS:
Other: Enhanced perioperative care protocol — See arm/group description
  Arms: Double Check enhanced perioperative care protocol

SUMMARY:
This multicenter open-label trial is designed to evaluate if the implementation of an enhanced peri-operative care protocol results in an optimal intraoperative condition of the patient and in a decrease in incidence of anastomotic leakage after colorectal resection as compared to current practice.

DETAILED DESCRIPTION:
Rationale Colorectal anastomotic leakage (CAL) remains a severe complication following surgery with a reported incidence of 3-19% worldwide. Recent research has identified several modifiable peri-operative CAL risk factors, suggesting that the intraoperative condition of the patient plays an important role in CAL development.

Objective To successfully implement an enhanced perioperative care protocol, focusing on optimizing the intraoperative condition of the patient to minimalize exposure to CAL risk factors. Secondly, to investigate whether implementation of this new guideline results in a better intraoperative condition and a decreased CAL rate as compared to current practice.

Study design An open-label multicenter design with historical cohort in nine participating hospitals.

Study population All adult patients that are scheduled for a colorectal resection with creation of a primary anastomosis.

Intervention An enhanced perioperative best practice protocol. The Double Check bundle exists out of interventions applicable without the introduction of new material to the operating room, on top of usual care. The protocol is based on the results of our previous large, multicenter, international observational cohort study (LekCheck study), systematic literature analyses, an inventory in current protocols on peri-operative care and expert opinion. Consensus is reached with colorectal surgeons from all participating centers. The final protocol was reviewed critically by experts in the field of colorectal surgery before implementation.

Comparison 1592 historical patients that were treated with standard practice (LekCheck study group). In addition the anastomotic leakage rates from the national registry of the period after the LekCheck study and before the start of the Double Check study will be used for comparison.

Endpoints Compliance to the study protocol, the patient's intraoperative condition and exposure to modifiable intraoperative risk factors, 30-day CAL and other postoperative complications according to Clavien-Dindo classification. Follow-up will be 90 days after colorectal resection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Bowel (small intestine/colon/rectal) resection with creation of a primary anastomosis
* Ability to give informed consent

Exclusion Criteria:

* The need for emergency surgery
* Scheduled operation concerning a reoperation for complications from recent surgery (within 3 months after the initial procedure).
* The inability to read or understand informed consent material

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2021-09-05 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of modifiable intraoperative CAL risk factors present during surgery as assessed by the DoubleCheck list | Intraoperative phase
  The primary outcome of the study is the intraoperative condition of the patient measured by the number of modifiable intraoperative CAL risk factors present in the patient.
  During the operation, the Double Check list will be completed.
  The list exists of 6 risk factors of interest:
  * Anemia: haemoglobin level < 7,5 (women) or < 8.0 (men) mmol/L
  * Hypothermia: temperature <36 degrees Celcius
  * Hyperglycemia: glucose level >10 mmol/L
  * Ue of vasopressor drugs: yes
  * Epidural analgesia
  * Incorrect antibiotic prophylaxis: not administered within 15-60 minutes prior to incision
  The number of risk factors present will be counted and a score of 0 to 6 will be given to each individual patient.

SECONDARY OUTCOMES:
Colorectal anastomotic leakage (CAL) | 30 days after surgery
  Defined as a grade B or C according to the ISREC classification
Postoperative complications | 30 days after surgery
  Defined as any adverse event occurring in the postoperative period until 30 days after surgery and graded according to the Dindo-Clavien classification
Postoperative mortality | 30 days after surgery
  Measured as rate of death at 30-day follow-up
Hospital Stay | 30 days after surgery
  Length of hospital and intensive care unit stay
Readmission | 30 days after surgery
  30-day readmission rate

CONTACTS AND LOCATIONS:
Locations (9):
- UZA, Antwerp, Belgium
- Netherlands (8):
  - Elkerliek, Helmond, Limburg
  - Maastricht UMC+, Maastricht, Limburg
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Bernhoven, Uden, North Brabant
  - Maxima Medisch Centrum, Veldhoven, North Brabant
  - Amsterdam UMC, Amsterdam, North Holland
  - Dijklander Ziekenhuis, Hoorn, North Holland
  - ZorgSaam, Terneuzen, Zeeland

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are/will be available upon request from dr. F. Daams
Time Frame: Upon request
Access Criteria: Upon request

REFERENCES:
- [Background] Huisman DE, Reudink M, van Rooijen SJ, Bootsma BT, van de Brug T, Stens J, Bleeker W, Stassen LPS, Jongen A, Feo CV, Targa S, Komen N, Kroon HM, Sammour T, Lagae EAGL, Talsma AK, Wegdam JA, de Vries Reilingh TS, van Wely B, van Hoogstraten MJ, Sonneveld DJA, Veltkamp SC, Verdaasdonk EGG, Roumen RMH, Slooter GD, Daams F. LekCheck: A Prospective Study to Identify Perioperative Modifiable Risk Factors for Anastomotic Leakage in Colorectal Surgery. Ann Surg. 2022 Jan 1;275(1):e189-e197. doi: 10.1097/SLA.0000000000003853. PMID 32511133
- [Background] van Rooijen SJ, Huisman D, Stuijvenberg M, Stens J, Roumen RMH, Daams F, Slooter GD. Intraoperative modifiable risk factors of colorectal anastomotic leakage: Why surgeons and anesthesiologists should act together. Int J Surg. 2016 Dec;36(Pt A):183-200. doi: 10.1016/j.ijsu.2016.09.098. Epub 2016 Oct 15. PMID 27756644
- [Derived] de Wit A, Bootsma BT, Huisman DE, Kazemier G, Daams F; Taskforce Anastomotic Leakage. Early detection and correction of preoperative anemia in patients undergoing colorectal surgery-a prospective study. Tech Coloproctol. 2025 Apr 5;29(1):92. doi: 10.1007/s10151-025-03131-5. PMID 40186755